CLINICAL TRIAL: NCT03299413
Title: Ulcerative Colitis Stem Cell Therapy
Brief Title: Use of Mesenchymal Stem Cells in Inflammatory Bowel Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hanan Jafar (Other)
Collaborators: Scientific Research Support fund (Unknown)
Responsible Party: Sponsor-Investigator, Hanan Jafar, DDS. MSc. PhD, University of Jordan
Organization: University of Jordan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBDUJCTC
Record Dates: First submitted 2017-09-27; First posted 2017-10-03 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Inflammatory Bowel Disease; Mesenchymal stem cells; Ulcerative colitis; Neutrophils
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wharton Jelly Mesenchymal stem cells (Experimental): Wharton Jelly Mesenchymal stem cells will be given as a cell suspension in aseptic buffered solution in disposable vials with no preservative agents. The cells will be injected every two weeks at a total of three doses, 120 million cells in 10mls divided on two IV boli for each dose
  Interventions: Biological: Wharton Jelly Mesenchymal stem cells

INTERVENTIONS:
Biological: Wharton Jelly Mesenchymal stem cells — Wharton Jelly Mesenchymal stem cells will be injected intravenously

SUMMARY:
Scientists hypothesize that directly or parentally injecting Mesenchymal stem cells (MSCs) to affected areas will have a positive impact through reducing or abolishing intestinal inflammation in part via inhibition of neutrophil Myeloperoxidase (MPOx) activity. Inhibiting MPOx should modify disease progression as well as reduce colitis associated cancer risk.

DETAILED DESCRIPTION:
Chronic inappropriate mucosal immune activation, due to aberrant host interactions with intestinal microbiota, is at the heart of inflammatory bowel disease (IBD) pathogenesis. Currently, there is no cure for IBD and mainstays of therapy are limited to non-cell specific immunosuppression/immunomodulation, antibiotics and surgery. Advanced ulcerative colitis patients cost approximately 10,000JD in therapy per year with 12.4% of patients presenting with rectal bleeding in Jordan being diagnosed with ulcerative colitis. The role of MSCs in immune modulation is well established in many diseases. However, the therapeutic potential of MSCs directly injected into the inflamed large intestine or parentally has not been fully investigated. Injected MSCs may modulate the IBD immune response particularly lymphoid T-cell and neutrophil activities. While a variety of immune cells contribute to the disease, increased neutrophil activity is associated with greater frequency and severity of active inflammation, as well as increased colitis associated cancer risk. MPOx can transform lipids and polyamines into reactive carbonyl species (RCS) capable of modifying proteins and DNA, altering cell signalling pathways. Finally, MPOx is reported as a useful tool in screening and risk stratification of human ulcerative colitis and colorectal cancer. Inhibiting MPOx in an accelerated preclinical mouse model did reduce incidence and tumor load resulting from gut inflammation. Additionally, in similar preclinical models others have reported that MSC transplantation reduces colitis severity and inflammatory markers including MPOx activity. Even in the absence of the well-known MSC T-cell immune modulation, disease activity indices and MPOx activity were reduced in these models. In addition to following traditional clinical outcomes, Reseachers will analyze gut immune responses, specifically neutrophil MPOx activity along with other IBD immune markers.

ELIGIBILITY:
Inclusion Criteria:

* Single/unmarried females or married females using two modalities of contraception for six months after completion of the study.
* Signed informed consent.
* Patients with previous diagnosis of ulcerative colitis (UC) or newly diagnosed UC based on endoscopic or histopathologic features
* Colitis of any activity

Exclusion Criteria:

* Mental disability that impedes adequate understanding of the study and of the associated procedures.
* Extensive severe toxic colitis requiring admission and IV steroids or biological treatment/surgery.
* Patients with previous colectomies.
* History of malignant disease.
* Pregnant or breastfeeding women.
* Presence of severe concomitant diseases such as chronic obstructive pulmonary disease, Diabetes Mellitus, Cardiovascular and other autoimmune diseases.
* Positive to one or more of the infectious disease panel

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-06-05 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 6 months
  Treatment adverse events are defined by any adverse event leading to hospitalization, organ failure or death

SECONDARY OUTCOMES:
Evaluation of the efficacy of the injected cells (Change from Baseline in partial mayo score) | 3 months
  Remission will be considered if reaches 0 points and response if the score diminishes. Endoscopy will be performed at 0 and 12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Cell Therapy Center, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided